CLINICAL TRIAL: NCT06945510
Title: A Multi-center Study to Evaluate the Economic and Clinical Impact of PCT Guided Antibiotics Use in Critically Ill Adult Patients in China.
Brief Title: PCT Guided Antibiotics Use in Critically Ill Adult Patients in China
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, YAN Shengtao, Deputy Director of the Emergency Department, China-Japan Friendship Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPLS-2173
Record Dates: First submitted 2025-04-14; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-10

CONDITIONS: Sepsis
Keywords: PCT
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCT group (Experimental): In the PCT group, clinicians will prescribe PCT tests every day for enrolled patients, with assigning a dedicated person monitoring the daily PCT results.
  Interventions: Device: PCT detection
- SOC group (No Intervention)

INTERVENTIONS:
Device: PCT detection — Clinicians will prescribe PCT tests every day for enrolled patients, with assigning a dedicated person monitoring the daily PCT results. Once the PCT <0.5 ng/ml or ΔPCT (drop from the peak value) >80%, the clinicians will receive a notification and will strictly adhere to guidelines and PCT values to adjust antibiotic prescriptions.
  Arms: PCT group

SUMMARY:
Procalcitonin (PCT) has been widely used in the diagnosis and treatment of bacterial infectious diseases in China. The investigators aim to establish an algorithm based on BRAHMS PCT (VIDAS PCT) for patients with severe infections or sepsis in the EICU to reduce antibiotic exposure and verify its validity in the reduction of antibiotic exposure, clinical outcomes and costs saving.

DETAILED DESCRIPTION:
This is a multi-center prospective study that will establish 9 centers. Based on preliminary on-site assessments, the centers will be grouped into two arms (SOC group and PCT group) according to their capacity for daily monitoring of PCT. Each center will enroll EICU patients with severe infections or sepsis who meet the inclusion and exclusion criteria. A total of 800 patients will be enrolled, with 400 in the PCT group and 400 in the SOC group. In the PCT group, clinicians will prescribe PCT tests every day for enrolled patients, with assigning a dedicated person monitoring the daily PCT results. Once the PCT <0.5 ng/ml or ΔPCT (drop from the peak value) >80%, the clinicians will receive a notification and will strictly adhere to guidelines and PCT values to adjust antibiotic prescriptions. The SOC group will not have any intervention regarding PCT prescriptions and antibiotic adjustments. The clinicians in the SOC group will prescribe PCT at routine frequency (usually once every 2-3 days or even longer) and adjust or discontinue antibiotics according to guidelines and their experiences. The primary and secondary endpoints will be evaluated in both groups. The primary endpoint is the total duration of antibiotic use. The secondary endpoints are the length of EICU stay and the total length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18
* Suspected or confirmed bacterial patients
* Stay EICU more than 3 days

Exclusion Criteria:

* age under 18 years;
* PCT concentration throughout the entire hospitalization less than 0.5 ng/ml ;
* known pregnancy; expected stay in the EICU less than 3 days;
* bone-marrow transplant or chemotherapy-induced neutropenia (<500 neutrophils per mL);
* infections for which long-term antibiotic treatment is strongly recommended (ie, infective endocarditis, osteoarticular infections, anterior mediastinitis after cardiac surgery, hepatic or cerebral abscesses, chronic prostatitis, or infection with Mycobacterium tuberculosis, Pneumocystis jirovecii, or Toxoplasma gondii);
* poor chance of survival, defined as a simplified acute physiology score (SAPS II) of more than 65 points at screening; and do-not-resuscitate orders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total duration of antibiotics use | From the day the patient was admitted to the EICU until the patient left the EICU, calculate how many days were antibiotics used.

SECONDARY OUTCOMES:
Total length of hospital stay (calculated in days) | The calculation starts from the first day the patient is admitted to the EICU and extends to the day the patient is discharged (including the possibility of the patient being transferred from the EICU to other departments).

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Austin PC. Informing power and sample size calculations when using inverse probability of treatment weighting using the propensity score. Stat Med. 2021 Nov 30;40(27):6150-6163. doi: 10.1002/sim.9176. Epub 2021 Sep 12. PMID 34510501
- [Background] Mewes JC, Pulia MS, Mansour MK, Broyles MR, Nguyen HB, Steuten LM. The cost impact of PCT-guided antibiotic stewardship versus usual care for hospitalised patients with suspected sepsis or lower respiratory tract infections in the US: A health economic model analysis. PLoS One. 2019 Apr 23;14(4):e0214222. doi: 10.1371/journal.pone.0214222. eCollection 2019. PMID 31013271
- [Background] Chow J, Markossian TW, Albarillo FS, Donahey EE, Bobay KL. Impact of a Procalcitonin-Based Protocol on Antibiotic Exposure and Costs in Critically Ill Patients. Crit Care Explor. 2021 Nov 9;3(11):e0571. doi: 10.1097/CCE.0000000000000571. eCollection 2021 Nov. PMID 34778793
- [Background] Hohn A, Balfer N, Heising B, Hertel S, Wiemer JC, Hochreiter M, Schroder S. Adherence to a procalcitonin-guided antibiotic treatment protocol in patients with severe sepsis and septic shock. Ann Intensive Care. 2018 Jun 4;8(1):68. doi: 10.1186/s13613-018-0415-5. PMID 29869120